CLINICAL TRIAL: NCT05628740
Title: A Phase 1, Two Part, Placebo-controlled, Single Dose Study in Healthy Volunteers and Multiple Dose Study in Patients With Refractory Chronic Cough to Assess the Safety, Tolerability, and PK of NTX-1175 Administered Via Nebulizer (NOC-100) and Dry Powder Inhaler (NOC-110)
Brief Title: Placebo-controlled, Single and Multiple Dose Study in Healthy Volunteers and Refractory Chronic Cough Patients to Assess the Safety, Tolerability, and Pharmacokinetics of Two Formulations of NTX-1175
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nocion Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: NOC110-C-102
Record Dates: First submitted 2022-11-02; First posted 2022-11-29 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2022-11

CONDITIONS: Refractory Chronic Cough
MeSH Terms: conditions — Chronic Cough

STUDY DESIGN:
Intervention Model Description: Part 1: randomized, double-blind, placebo-controlled, 3-period crossover, and 1-period parallel study.
  Part 2: randomized, double-blind, placebo-controlled, multiple-dose, parallel-design.
Who Masked: Participant, Investigator
Masking Description: A computerized randomization scheme for Part 1 and Part 2 will be created by a blinded study statistician and it shall be considered blinded per the following: The randomization is available only to the unblinded Clinic pharmacy staff who are preparing the study drug and who will not be involved in any other aspect of the study including administration of the study drug. The randomization scheme will not be made available to the Sponsor, study participants, or members of the staff responsible for the monitoring and evaluation of safety assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part 1-Period 1-Treatment A (Experimental): 3 mg NOC-100 (via nebulizer)
  Interventions: Drug: 3 mg NOC-100 (via nebulizer)
- Part 1-Periods 2 through 4 -Treatment B (Placebo Comparator): 1 mg NOC-110 DPI (1 capsule)
  Interventions: Drug: 1 mg NOC-110 (via DPI) [1x 1 mg capsule]
- Part 1-Periods 2 through 4 - Treatment C (Placebo Comparator): 3mg NOC-110 DPI (1 capsule)
  Interventions: Drug: 3 mg NOC-110 (via DPI)
- Part 1-Periods 2 through 4- Placebo (Placebo Comparator): Placebo (1 capsule)
  Interventions: Drug: Placebo (via DPI)
- Part 1-Period 5- Treatment D (Placebo Comparator): 6mg NOC-110 DPI (2 capsules)
  Interventions: Drug: 6 mg NOC-110 (via DPI)
- Part 1-Period 5- Placebo (Placebo Comparator): Placebo (2 capsules)
  Interventions: Drug: Placebo (via DPI) [2x Placebo capsules]
- Part 2- Active (Placebo Comparator): 6mg NOC-110 DPI (2 capsules)
  Interventions: Drug: 6 mg NOC-110 (via DPI)
- Part 2- Placebo (Placebo Comparator): Placebo DPI (2 capsules)
  Interventions: Drug: Placebo (via DPI) [2x Placebo capsules]

INTERVENTIONS:
Drug: 3 mg NOC-100 (via nebulizer) — Participants determined to be eligible for Part 1 of the study will be enrolled and will be assigned to receive a single dose of the reference nebulizer treatment of NOC 100 at 3 mg (Treatment A) in Period 1
  Arms: Part 1-Period 1-Treatment A
Drug: 1 mg NOC-110 (via DPI) [1x 1 mg capsule] — Participants will be randomized to receive single doses of 1 mg NOC-110 (via DPI) in a crossover fashion according to a prespecified randomization schedule
  Arms: Part 1-Periods 2 through 4 -Treatment B
Drug: 3 mg NOC-110 (via DPI) — Participants will be randomized to receive single doses of 3 mg NOC-110 (via DPI) in a crossover fashion according to a prespecified randomization schedule
  Arms: Part 1-Periods 2 through 4 - Treatment C
Drug: Placebo (via DPI) — Participants will be randomized to receive single doses of placebo via capsule in a crossover fashion according to a prespecified randomization schedule
  Arms: Part 1-Periods 2 through 4- Placebo
Drug: 6 mg NOC-110 (via DPI) — Participants will be randomized to receive single doses of 6 mg NOC-110 via DPI in a parallel fashion according to a prespecified randomization schedule
  Arms: Part 1-Period 5- Treatment D; Part 2- Active
Drug: Placebo (via DPI) [2x Placebo capsules] — Participants will be randomized to receive single doses of Placebo (via DPI) [2x Placebo capsules] in a parallel fashion according to a prespecified randomization schedule
  Arms: Part 1-Period 5- Placebo; Part 2- Placebo

SUMMARY:
Part 1 will evaluate the safety, tolerability and PK of single doses of three dose levels of NTX-1175 drug substance administered by dry powder inhaler (NOC-110) compared to a single dose reference nebulizer (NOC-100) treatment in healthy participants.

Part 2 will evaluate the safety, tolerability and PK of multiple doses of NTX-1175 drug substance administered by dry powder inhaler (NOC-110) to participants with refractory chronic cough. Part 2 will also evaluate the treatment effect of multiple doses of one dose level of NTX-1175 drug substance administered by dry powder inhaler (NOC-110).

DETAILED DESCRIPTION:
Part 1 is a randomized, double-blinded 3 period crossover and 1 period parallel study of single dose administration of NOC-110 via dry powder inhaler, preceded by a reference period of NOC-100 administered via nebulizer. A total of 12 healthy participants will be enrolled to ensure that 9 participants complete this part of study.

Part 2 is a randomized, double-blinded, placebo-controlled, multiple-dose, parallel design study in patients with refractory chronic cough. A total of 12 participants will be enrolled to ensure that 8 participants complete this part of study.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria to be eligible for participation in the study:

1. Male or female participants between the ages of 18 to 65 years, inclusive, at the time of screening (Part 1) and between the ages of 18 to 85 years, inclusive, at the time of screening (Part 2).
2. Has had rCC diagnosis for ≥ 12 months (Part 2) prior to screening.
3. Awake-cough frequency of ≥20 per hour (average) at Screening (Part 2).
4. Score of ≥40 mm on the Cough Severity Visual Analog Scale (VAS) at Screening (Part 2).
5. Chest radiograph or CT thorax within the last 60 months not demonstrating any abnormality considered to be significantly contributing to the rCC. (Part 2)
6. Body mass index (BMI) ≥19.0 and ≤32.0 kg/m2, inclusive, at Screening.
7. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <2 x upper limit of normal (ULN); alkaline phosphatase (ALP) and bilirubin ≤1.5 x ULN (isolated bilirubin >1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
8. Creatinine clearance ≥50 mL/min.
9. Must be fully SARS-CoV-2 vaccinated.
10. Must be SARS-CoV-2 negative via rapid antigen testing or polymerase chain reaction (PCR) test at Screening and PCR at Check-in Day -1.
11. In the Investigator's opinion, has no clinically significant disease and/or clinically significant abnormal laboratory values as determined by the Investigator based on medical history, physical examination, or laboratory evaluations conducted at the screening visit or on admission to the clinical research unit.

Exclusion Criteria:

Participants who meet any one of the following criteria will be deemed ineligible for participation in the study:

1. Is found to have positive test for SARS-CoV-2 at Screening or Check-in Day -1, whether or not this was accompanied by the clinical symptoms of COVID-19.
2. Current smoker or individuals who have given up smoking within the past 6 months prior to screening, or those with >20 pack-year smoking history (Part 2)
3. Current diagnosis of chronic obstructive pulmonary disease (COPD), bronchiectasis, unexplained pulmonary fibrosis, or asthma (Part 2).
4. History or presence of alcohol or drug use disorder, per Diagnostic and Statistical Manual of Mental Disorders, fifth edition (DSM-5), within the past 2 years prior to screening.
5. Current opiate/opioid use in the past 7 days prior to screening, or medical history of opiate/opioid use disorder.
6. Unable to refrain from the use of:

   1. Gabapentin, pregabalin, and/or amitryptline or other tricyclics within 4 weeks prior to screening and throughout the study (Part 2)
   2. Chronic, systemic corticosteroid use within 4 weeks prior to screening and throughout the study (Part 2).
   3. Inhalers including long-acting and short acting beta 2-agonists (LABA and SABA), and inhaled corticosteroids (ICS) within 8 weeks prior to screening and throughout the study.
   4. Lidocaine or related compounds of any form within 14 days prior to screening and throughout the study (Part 2).
   5. Medication or remedies to aid sleeping 14 days prior to screening and throughout the study (Part 2).
   6. Angiotensin-converting enzyme (ACE)-inhibitor within 12 weeks prior to screening and throughout the study (Part 2).
   7. Antitussives 7 days prior to screening and throughout the study (Part 2).
   8. Speech and language therapy for rCC within 4 weeks prior to screening and throughout the study (Part 2).
   9. Food and beverages containing alcohol for 24 hours prior to screening (Part 2).
7. History or presence of cardiac dysfunction including arrhythmia, bundle branch block; Wolff Parkinson White syndrome, recent thromboembolic event, prolonged PR (≥220 msec), QRS (≥120 msec), QTcF interval (≥450 msec [males] or ≥470 msec [females]) or has ECG findings deemed abnormal with clinical significance by the Investigator or designee at Screening.
8. Positive results at Screening for HIV, HBsAg, or HCV (participants successfully treated for HCV may be permitted at the discretion of the Investigator).
9. Supine blood pressure is less than 90/40 mmHg or greater than 140/90 mmHg (Part 1), or greater than 160/95 mmHg (Part 2) at Screening. Vital signs may be repeated twice.
10. Supine heart rate is lower than 40 beats per minute (bpm) or higher than 99 bpm at Screening. Vital signs may be repeated twice.
11. History of asthma or COPD (Part 1).
12. Forced expiratory volume in 1 second/ forced vital capacity (FEV1/FVC) < lower limit of normal (LLN) per Global Lung Health Initiative normative dataset at Screening.
13. Had symptoms of any significant acute illness, including symptoms of COVID-19 within 30 days before the start of the study (time of first dose), as determined by the Investigator.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2022-10-25 (Actual)

PRIMARY OUTCOMES:
Number and severity of Treatment Emergent Adverse Events (TEAEs) following single doses of NOC-110 or placebo administered with a DPI | Part 1- Screening through Day 23
  To evaluate the safety and tolerability of single doses of three dose levels of NTX-1175 drug substance administered by DPI (Drug Product NOC-110) compared to a single dose reference nebulizer treatment (Drug Product NOC-100) in healthy participants, number and severity of TEAEs following single doses of NOC-110 or placebo administered with a DPI compared to a reference period administration of NOC 100 via a nebulizer in healthy adult participants will be reported.
Number and severity of TEAE following repeat doses of NOC 110 compared to placebo in participants with chronic cough. | Part 2- Screening through Day 12
  To evaluate the safety and tolerability of multiple doses of NOC-110 administered by DPI to participants with refractory chronic cough (rCC), number and severity of TEAE following repeat doses of NOC 110 compared to placebo in participants with chronic cough will be reported.

SECONDARY OUTCOMES:
Peak plasma concentration (Cmax) of single doses of three dose levels of NOC-110 administered by DPI compared to a single dose reference nebulizer treatment (NOC-100) in healthy participants. | Part 1- Day 1, Day 5, Day 9, Day 13 and Day 17
  PK parameters for plasma NTX-1175:
  Cmax
The time to reach maximum observed concentration (Tmax) of single doses of three dose levels of NOC-110 administered by DPI compared to a single dose reference nebulizer treatment (NOC-100) in healthy participants. | Part 1- Day 1, Day 5, Day 9, Day 13 and Day 17
  PK parameters for plasma NTX-1175:
  Tmax
The area under the concentration-time (AUC) curve of single doses of three dose levels of NOC-110 compared to a single dose reference nebulizer treatment in healthy participants. | Part 1- Day 1, Day 5, Day 9, Day 13 and Day 17
  PK parameters for plasma NTX-1175:
  AUC [time 0 to the last observed non-zero concentration (t) (AUC0-t), time 0 to Hour 24 (AUC0-24), time 0 extrapolated to infinity (AUC0-inf), percent of AUC0 inf extrapolated (AUC%extrap)]
The time of the last measurable concentration (Tlast) of single doses of three dose levels of NOC-110 administered by DPI compared to a single dose reference nebulizer treatment (NOC-100) in healthy participants. | Part 1- Day 1, Day 5, Day 9, Day 13 and Day 17
  PK parameters for plasma NTX-1175:
  Tlast
The apparent terminal elimination half-life (t½) of single doses of three dose levels of NOC-110 administered by DPI compared to a single dose reference nebulizer treatment (NOC-100) in healthy participants. | Part 1- Day 1, Day 5, Day 9, Day 13 and Day 17
  PK parameters for plasma NTX-1175:
  t½
The apparent terminal elimination rate constant (Kel) of single doses of three dose levels of NOC-110 administered by DPI compared to a single dose reference nebulizer treatment (NOC-100) in healthy participants. | Part 1- Day 1, Day 5, Day 9, Day 13 and Day 17
  PK parameters for plasma NTX-1175:
  Kel
The Cmax of multiple doses of NOC 110 administered by DPI to participants with rCC. | Part 2- Day 1, Day 5
  PK parameters for plasma NTX-1175:
  Cmax and maximum observed concentration at steady-state (Cmax, ss)
The Tmax of multiple doses of NOC 110 administered by DPI to participants with rCC. | Part 2- Day 1, Day 5
  PK parameters for plasma NTX-1175:
  Tmax, time to reach Cmax,ss (Tmax,ss)
The AUC of multiple doses of NOC 110 administered by DPI to participants with rCC. | Part 2- Day 1, Day 5
  PK parameters for plasma NTX-1175:
  AUC0-t AUC0-inf AUC%extrap
The Tlast of multiple doses of NOC 110 administered by DPI to participants with rCC. | Part 2- Day 1, Day 5
  PK parameters for plasma NTX-1175:
  Tlast
The t½ of multiple doses of NOC 110 administered by DPI to participants with rCC. | Part 2- Day 1, Day 5
  PK parameters for plasma NTX-1175:
  t½
The Kel multiple doses of NOC 110 administered by DPI to participants with rCC. | Part 2- Day 1, Day 5
  PK parameters for plasma NTX-1175:
  Kel
The concentration observed at the end of the dosing interval (Ctrough) of multiple doses of NOC 110 administered by DPI to participants with rCC. | Part 2- Days 2 to 4
  PK parameters for plasma NTX-1175:
  Ctrough
The minimum observed non zero concentration between dose time and dose time + dosing interval (tau) (min,ss,) of multiple doses of NOC 110 administered by DPI to participants with rCC. | Part 2- Day 5
  PK parameters for plasma NTX-1175:
  Cmin,ss
The area under the concentration-time curve during a dosing interval (tau), at steady state (AUCtau) of multiple doses of NOC 110 administered by DPI to participants with rCC. | Part 2- Day 5
  PK parameters for plasma NTX-1175:
  AUCtau
The average concentration during a dosing interval, at steady state (Cavg,ss) of multiple doses of NOC 110 administered by DPI to participants with rCC. | Part 2- Day 5
  PK parameters for plasma NTX-1175:
  Cavg,ss
The accumulation (R) of multiple doses of NOC 110 administered by DPI to participants with rCC. | Part 2- Day 5
  PK parameters for plasma NTX-1175:
  R
Awake-coughs per hour in participants with rCC | Part 2- Screening, Day -1, Day 1, Day 3 and Day 5
  The treatment effect of multiple doses of one dose level of NOC-110 administered by DPI, as determined by awake-coughs per hour in participants with rCC.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Silber, MD, Study Director — Nocion Therapeutics, Inc.
Locations (3):
- United States (3):
  - Celerion, Phoenix, Arizona
  - Clinical Site Partners, Leesburg, Florida
  - Clinical Site Partners, Winter Park, Florida